CLINICAL TRIAL: NCT06416111
Title: Comparison of Infraclavicular Brachial Plexus Block and Local Anesthesia in Arteriovenous Fistula Surgeries and Their Effects on Tissue Oxygen Saturation With Near-infrared Spectroscopy
Brief Title: Comparison of Infraclavicular Brachial Plexus Block and Local Anesthesia in Arteriovenous Fistula Surgeries and Their Effects on Tissue Oxygen Saturation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Hija Yazıcıoğlu, Prof.MD, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Tissue Oxygen Saturation
Record Dates: First submitted 2024-04-26; First posted 2024-05-16 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Renal Disease, Chronic
Keywords: arteriovenous fistula operation; Infraclavicular nerve block; Near-infrared spectroscopy (NIRS); local anesthesia
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Bupivacaine; Prilocaine

STUDY DESIGN:
Intervention Model Description: NIRS probes will be placed on the thenar, antecubital regions of both hands and arms .The preoperative observed values and data of every 5 minutes during the operation will be recorded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local group(Group L) (Active Comparator): Local infiltrative anesthesia will be applied with 15 ml 2% prilocaine for Local group patients.Before surgery, NIRS probes will be placed on the thenar, antecubital regions of both hands and arms .The peripheral regional oxygen saturation values will be recorded preoperatively and every 5 minutes during the operation.
  Surgeon and patient satisfaction will be evaluated by 5 Point Likert Scale (worst: 1 point, best: 5 points) at the end of the surgery.
  Interventions: Device: NIRS; Drug: Prilocaine
- Block group(Group B) (Active Comparator): For Block group patients, 30 ml 0.25% bupivacaine will be applied with Infraclavicular approach around brachial plexus with inplane technique.The effect of the peripheral nerve block will be evaluated with 10-minute intervals until regional anesthesia is achieved.Sensory block will be evaluated with the "Pinprick Test" and motor block with the "Modified Bromage Scale". For patients who underwent a block, Grade 2 on the "Pinprick Test" and Grade 3 on the "Modified Bromage Scale" were considered suitable anesthesia conditions for the operation. Before surgery, NIRS probes will be placed on the thenar, antecubital regions of both hands and arms .The peripheral regional oxygen saturation values will be recorded preoperatively and every 5 minutes during the operation.
  Surgeon and patient satisfaction will be evaluated by 5 Point Likert Scale (worst: 1 point, best: 5 points) at the end of the surgery.
  Interventions: Device: NIRS; Other: Pinprick Test; Other: Modified Bromage Scale; Drug: Bupivacaine

INTERVENTIONS:
Device: NIRS — Near Infra-Red Spectroscopy (NIRS) is a non-invasive monitoring modality which measures regional tissue oxygenation defined as percentage (%).
Other: Pinprick Test — With the pinprick test, the practitioner gently touches the skin with the pin and asks the patient whether it feels sharp or blunt .Test begins distally and then move proximally (aiming to test each dermatome and each main nerve).
  Assessment of sensorial blockade uses 3 grade system. Grade 0.Sharp pain Grade 1.Analgesia ,numbness Grade 2.Anesthesia ,no feeling
  Arms: Block group(Group B)
Other: Modified Bromage Scale — Assessment of motor blockade uses 4 point Modified Bromage Score. 0.Normal motor function with full extension and flexion of elbow, wrist and fingers
  1. Decreased motor strengths with ability to full flexion elbow and move fingers but inability to raise arm
  2. More decreased motor strengths with inability to move elbow but ability to move fingers 3.Complete motor block with inability to move elbow, wrist, and fingers.
  Arms: Block group(Group B)
Drug: Bupivacaine — Bupivacaine is a potent local anesthetic with unique characteristics from the amide group of local anesthetics.
  Other Names: Marcaine; Sensorcaine
  Arms: Block group(Group B)
Drug: Prilocaine — Prilocaine is an amide local anesthetic secondary amine with an intermediate length of duration and quick onset of action.
  Other Names: Citanest; Propitocaine; Xylonest
  Arms: Local group(Group L)

SUMMARY:
In arteriovenous fistula surgery, the effect of infraclavicular brachial plexus block and local anesthesia on tissue oxygenation and the effect of primary patency of the AV fistula is intended to research.

DETAILED DESCRIPTION:
It is planned to include patients who are American Society of Anesthesiologists (ASA) III and between the ages of 18-80 who will undergo arteriovenous fistula surgery in the research population.In our study, patients who come to the operating room for arteriovenous fistula operation will be randomly divided into two groups.Patients who undergo simple randomization with coin toss method will be assigned to one of two groups: group Local infiltrative anesthesia (Local) and group infraclavicular brachial plexus block with 0.25% bupivacaine (Block). Local infiltrative anesthesia will be applied with 15 ml 2% prilocaine for group Local patients.For Group Block patients, 30 ml 0.25% bupivacaine will be applied with Infraclavicular approach around brachial plexus with inplane technique.Before the start of surgery, NIRS probes will be placed on the thenar ,antecubital regions of both hands and arms .The preoperative observed values and data of every 5 minutes during the operation will be recorded .

ELIGIBILITY:
Inclusion Criteria:

* ASA III
* 18-80 years old
* arteriovenous fistula operation

Exclusion Criteria:

* disabled patients
* mentally retarded
* patients with coagulopathy
* hemoglobinopathy
* patients with infection in the infraclavicular area
* local anesthetic history
* peripheral neuropathy
* peripheral arterial occlusion
* failed peripheral nerve block

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-22 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
tissue oxygenation | beginning and every 5 minutes till the end of surgery
  To compare the effects of infraclavicular brachial plexus block and local infiltrative anesthesia on tissue oxygenation during arteriovenous fistula (AVF) surgeries.
  Near Infra-Red Spectroscopy (NIRS) is a non-invasive monitoring modality which measures regional tissue oxygenation defined as percentage (%).Before surgery, NIRS probes will be placed on the thenar, antecubital regions of both hands and arms .
primary patency of the arteriovenous fistula | 1 month after the operation
  To compare the effects of infraclavicular brachial plexus block and local infiltrative anesthesia on the primary patency of the arteriovenous fistula

SECONDARY OUTCOMES:
5 Point Likert Scale | at the end of the operation
  Surgeon and patient satisfaction will be evaluated by 5 Point Likert Scale at the end of surgery.
  1 point:Dissatisfaction; 5 point:Fully satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Hija Yazıcıoğlu, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No